CLINICAL TRIAL: NCT04119908
Title: Interest of Sublingual Videomicroscopy for the Prediction of Bleeding in Von Willebrand Disease and Other Constitutional Haemorrhagic Diseases
Brief Title: Videomicroscopy for the Prediction of Bleeding in Constitutional Haemorrhagic Diseases
Acronym: VIDEO-BLEED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019_05; 2019-A01601-56 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Von Willebrand Diseases; Glanzmann Thrombasthenia
Keywords: constitutional haemorrhagic diseases, Videomicroscopy, prediction, bleeding; Videomicroscopy; prediction; bleeding
MeSH Terms: conditions — von Willebrand Diseases; Thrombasthenia; Hemorrhage | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with haemorrhagic disease (Experimental): Patients with von Willebrand disease or Patients with Glanzmann Thrombasthenia
  Interventions: Device: Sublingual videomicroscopy; Biological: blood sample
- Control group (Other): Patients with moderate or severe hemophilia A or women carrying the hemophilia gene
  Interventions: Device: Sublingual videomicroscopy

INTERVENTIONS:
Device: Sublingual videomicroscopy — Measurement of sublingual capillary density by video microscopy
Biological: blood sample — Collection of citrate tubes of 5 mL at baseline and at 36 months
  Arms: Patients with haemorrhagic disease

SUMMARY:
In Willebrand disease, there is currently no test available to identify non-invasively patients with a high risk of bleeding from angiodysplasias The study propose to use a sublingual capillary bed analysis by video-microscopy, a sensitive, reproducible and non-invasive technique, to assess whether sublingual capillary density is predictive of hemorrhagic risk for patients with von Willebrand disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with a significant form of von Willebrand disease (according to the inclusion criteria of the Willebrand Disease French Reference Center), a Glanzmann Thrombasthenia, a moderate to severe Haemophilia A or a woman carrying the hemophilia gene
* Social insured patient

Exclusion Criteria:

* Minor patient
* Refusal of consent
* Person benefiting from a system of legal protection
* Pregnant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2028-05-24 (Estimated); Study Completion 2028-05-24 (Estimated)

PRIMARY OUTCOMES:
area under the ROC curve from Sublingual capillary density to inclusion for the event "existence of at least a clinically significant haemorrhage" | at 3 years

SECONDARY OUTCOMES:
Sublingual capillary density | At baseline
  To compare the sublingual capillary density of patients with von Willebrand disease to that of 3 other groups of patients:
  * with a severe form of hemophilia A
  * with a moderate form of hemophilia A
  * women carrying the hemophilia gene
qualitative abnormalities of sublingual capillaries (capillary haemorrhage, capillary dystrophy) | At baseline and at 3 years
  presence or absence of qualitative abnormalities
delta of Sublingual capillary density increase | between inclusion and end of study (at 3 years)
ISTH-BAT haemorrhagic score (International Society on Thrombosis and Hemostasis - Bleeding Assessment Tool) | At baseline, at 3 years
  ISTH-BAT is a questionnaire minimum score ranges from 0 to 10 whereas maximum score ranges from 20 to 30
delta of increase of ISTH-BAT haemorrhagic score | between inclusion and end of study (at 3 years)
  ISTH-BAT is a questionnaire minimum score ranges from 0 to 10 whereas maximum score ranges from 20 to 30
plasma levels of proangiogenic markers | at inclusion and end-of-study visits(at 3 years)
  dosage of angiopoietin-1, angiopoetin-2 (pg/mL) measured by ELISA
plasma levels of galectine | at inclusion and end-of-study visits(at 3 years)
  galectin-1 and galectin-3 measured by ELISA
plasma levels of VEGF | at inclusion and end-of-study visits(at 3 years)
  Concentration (pg/ml) of Vascular Endothelial Growth Factor (VEGF) in blood measured by ELISA
delta of increase in plasma levels of all proangiogenic markers | At inclusion and end of study (at 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Rauch, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU de Lille, Lille, Nord, France